CLINICAL TRIAL: NCT00476086
Title: A Phase II Study of Oxaliplatin and Gemcitabine Followed by Radiation Therapy in the Management of Mixed Mullerian Tumors of the Uterus
Brief Title: Oxaliplatin and Gemcitabine Followed by Radiation Therapy in the Management of Mixed Mullerian Tumors of the Uterus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Sanofi (Industry); Brigham and Women's Hospital (Other); Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Susana M. Campos, MD, Medical Oncologist, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-063
Record Dates: First submitted 2007-05-17; First posted 2007-05-21 (Estimated); Results first posted 2016-04-13 (Estimated); Last update posted 2018-08-24 (Actual); Status verified 2018-07

CONDITIONS: Mixed Mullerian Tumors of the Uterus
Keywords: oxaliplatin; gemcitabine; MMMT
MeSH Terms: interventions — Gemcitabine; Oxaliplatin; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Oxaliplatin/ Gemcitabine Then Radiation (Experimental): Patients rcvd IV chemotherapy on days 1 and 15 of a 4-week cycle: gemcitabine 1000 mg/m2 and oxaliplatin 65 mg/m2 for up to 3 cycles. Two dose reductions per study drug were permitted. On study, chemotherapy was followed by radiation therapy (RT) within 4-6 weeks of last chemotherapy. RT regimen was tumor-volume directed.
  Interventions: Drug: Gemcitabine; Drug: Oxaliplatin; Radiation: Radiation

INTERVENTIONS:
Drug: Gemcitabine
  Other Names: Gemzar
Drug: Oxaliplatin
  Other Names: Eloxatin
Radiation: Radiation

SUMMARY:
The purpose of this research study is to determine the feasibility and safety of giving the combination of oxaliplatin and gemcitabine followed by radiation therapy and to learn whether or not this drug combined with radiation therapy works in treating women with Mullerian tumors of the uterus.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary To determine the feasibility of dual modality therapy described as cytotoxic therapy followed by radiation therapy for the management of Malignant Mixed Mullerian Tumors (MMMTs).

Secondary

* To describe the response rate by Response Evaluation Criteria in Solid Tumors

STATISTICAL DESIGN:

This study used a two-stage design to evaluate feasibility of oxaliplatin and gemcitabine prior to radiation therapy defined as completing 3 cycles of chemotherapy. The null and alternative therapy completion rates were 25% and 50%. If 3 or more participants enrolled in the stage one cohort (n=9 participants) complete therapy than accrual would proceed to stage two (n=15 participants). If therapy was completed by at least 10 participants in the final set of 24 evaluable participants then this regimen would be deemed worthy of further study. This design had 80% power given one-sided type I error of 5% with the probability of stopping early 0.60.

ELIGIBILITY:
Inclusion Criteria:

* Surgically staged and histologically confirmed diagnosis of MMMT
* 18 years of age or older
* ECOG Performance Score of 0-2
* Adequate bone marrow function
* Adequate renal function
* Adequate hepatic function
* Patients must be recovered from both the acute and late effects of any prior surgery

Exclusion Criteria:

* Patients with an active infection
* Patients with CNS metastases
* History of prior malignancy within the past 5 years except curatively treated basal cell carcinoma of the skin, or cervical intraepithelial neoplasia
* Known hypersensitivity to any of the components of oxaliplatin or gemcitabine
* Prior radiation to the pelvis
* Patients who are receiving concurrent investigational therapy or who have received investigational therapy within 30 days
* Peripheral neuropathy greater or equal to Grade 2
* Stage IV visceral disease (lung and liver metastases at presentation)
* Any other medical condition, including mental illness or substance abuse, deemed by the investigator to be likely to interfere with a patient's ability to sign informed consent
* Known HIV or Hepatitis B or C (active, previously treated or both)
* Pregnant or breast feeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-08; Primary Completion 2012-03 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susana Campos, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 20 participants were enrolled between May 2007 and August 2011.
Groups:
- Oxaliplatin/ Gemcitabine Then Radiation: Patients received IV chemotherapy on days 1 and 15 of a 4-week cycle: gemcitabine 1000 mg/m2 and oxaliplatin 65 mg/m2 for up to 3 cycles. Two dose reductions per study drug were permitted. On study, chemotherapy was followed by radiation therapy (RT) within 4-6 weeks of last chemotherapy. RT regimen was tumor-volume directed.
Period: Overall Study
Arm/Group | Oxaliplatin/ Gemcitabine Then Radiation
Started | 20
Received Chemotherapy | 19
Received Radiation | 15
Completed | 15
Not Completed | 5
Not completed — Alternative therapy | 1
Not completed — Progressive Disease | 4

BASELINE CHARACTERISTICS:
Population: The baseline population is comprised of all enrolled patients.
Groups:
- Oxaliplatin/ Gemcitabine Then Radiation: Patients rcvd IV chemotherapy on days 1 and 15 of a 4-week cycle: gemcitabine 1000 mg/m2 and oxaliplatin 65 mg/m2 for up to 3 cycles. Two dose reductions per study drug were permitted. On study, chemotherapy was followed by radiation therapy (RT) within 4-6 weeks of last chemotherapy. RT regimen was tumor-volume directed.
  on
Arm/Group | Oxaliplatin/ Gemcitabine Then Radiation
Number analyzed (Participants) | 20
Age, Continuous [Mean (Full Range); unit: years] | 63 [49 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Chemotherapy Completion Rate
Description: Feasibility in this study was based on the chemotherapy regimen. The chemotherapy completion rate is defined as the percentage of patients who complete 3 cycles of oxaliplatin and gemcitabine chemotherapy prior to radiation therapy.
Time Frame: 3 cycles of chemotherapy which approximates 3 months given the 28-day cycle
Population: The analysis dataset is comprised of all participants who started chemotherapy.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Oxaliplatin/ Gemcitabine Then Radiation
Number analyzed (Participants) | 19
percentage of participants | 100 [85 to 100]

2. Secondary Outcome: Radiation Therapy Completion Rate
Description: Disease was evaluated radiologically at baseline and every X cycles on treatment; Treatment continued if radiological exam showed no progressive disease
Time Frame: Radiation therapy was within 4-6 weeks of last chemotherapy dose. Participants received up to 5 weeks of radiation therapy.
Population: The analysis dataset is comprised of all participants who started chemotherapy.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Oxaliplatin/ Gemcitabine Then Radiation
Number analyzed (Participants) | 19
percentage of participants | 79 [58 to 92]

ADVERSE EVENTS:
Time Frame: Assessed each cycle of chemotherapy and week of radiation therapy from time of first dose and up to day 30 post-treatment. Participants received a median of 3 cycles (1 cycle = 4 weeks) of chemotherapy and 5 weeks of radiation therapy.
Description: Maximum grade toxicity by type was first calculated within two subsets reflecting either adverse events with treatment-attribution of possibly, probably or definitely.related to chemotherapy or radiation therapy Serious and Other AEs were defined as grades 3-5 and grades 1-2, respectively, per CTCAEv3. (Evaluation excludes untreated participants.)
Groups:
- Oxaliplatin/ Gemcitabine: Patients rcvd IV chemotherapy on days 1 and 15 of a 4-week cycle: gemcitabine 1000 mg/m2 and oxaliplatin 65 mg/m2 for up to 3 cycles. Two dose reductions per study drug were permitted.
- Radiation: On study, chemotherapy was followed by radiation therapy (RT) within 4-6 weeks of last chemotherapy. RT regimen was tumor-volume directed.
Arm/Group | Oxaliplatin/ Gemcitabine | Radiation
Serious Adverse Events (participants affected / at risk) | 2/19 | 2/15
Other Adverse Events (participants affected / at risk) | 15/19 | 14/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oxaliplatin/ Gemcitabine (N=19) | Radiation (N=15)
Infection Gr0-2 neut, colon (Infections and infestations) | 1 | 0
ALT, SGPT (Investigations) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oxaliplatin/ Gemcitabine (N=19) | Radiation (N=15)
Abdomen, pain (Gastrointestinal disorders) | 0 | 3
Allergic reaction (Immune system disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 0
ALT, SGPT (Investigations) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 2
Anxiety (Psychiatric disorders) | 1 | 0
AST, SGOT (Investigations) | 1 | 0
Back, pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 8 | 3
Constitutional, other (General disorders) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 2 | 11
Dizziness (Nervous system disorders) | 1 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 3 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Edema limb (General disorders) | 0 | 1
Extremity-limb, pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Fatigue (General disorders) | 14 | 9
Fever w/o neutropenia (General disorders) | 1 | 0
Flushing (Vascular disorders) | 1 | 1
GI-other (Gastrointestinal disorders) | 2 | 1
Head/headache (Nervous system disorders) | 1 | 0
Hemoglobin (Blood and lymphatic system disorders) | 1 | 0
Hemorrhoids (Gastrointestinal disorders) | 0 | 3
Hot flashes (Vascular disorders) | 1 | 1
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 0
Infection w/ gr3-4 neut, anal/perianal (Infections and infestations) | 1 | 0
Infection-other (Infections and infestations) | 0 | 1
Injection site reaction (General disorders) | 3 | 0
Joint, pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Leukocytes (Investigations) | 2 | 1
Muscle, pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Musculoskeletal/soft tissue-other (Musculoskeletal and connective tissue disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 10 | 6
Neurologic-other (Nervous system disorders) | 12 | 5
Neuropathy-sensory (Nervous system disorders) | 9 | 1
Neutrophils (Investigations) | 0 | 2
Pain NOS (General disorders) | 1 | 0
Pain-other (General disorders) | 1 | 1
Platelets (Investigations) | 2 | 0
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1 | 0
Radiation dermatitis (Injury, poisoning and procedural complications) | 0 | 5
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 | 2
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 2 | 0
Rectum, pain (Gastrointestinal disorders) | 0 | 1
Rigors/chills (General disorders) | 1 | 0
Skin, pain (Skin and subcutaneous tissue disorders) | 1 | 2
Skin-other (Skin and subcutaneous tissue disorders) | 2 | 0
Taste disturbance (Nervous system disorders) | 2 | 0
Urinary frequency/urgency (Renal and urinary disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 4 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No